CLINICAL TRIAL: NCT01314157
Title: Evaluation of Isostretching Effects in Patients With Mechanical and Postural
Brief Title: Evaluation of Isostretching Effects in Patients With Mechanical and Postural Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Erika Rosangela Alves Prado, Mestra em Ciências da Saúde Aplicada a Medicina Reumatológica, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Prado
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; pain; incapacity; life quality; rehabilitation
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Intervention Model Description: Alocados de forma cega para o grupo de intervenção: 27 pacientes com diagnóstico de lombalgia crônica realizaram o Isostretching e uso de diclofenaco em caso de dor e grupo controle:27 pacientes com lombalgia crônica sem atividade física com uso apenas de diclofenaco em caso dedor Todos foram submetidos à avaliação inicial (T0), com 20 dias (T20) e com 45 dias (T45), por um avaliador cego. Os pacientes foram instruídos nos dois grupos, pelo médico, a utilizar o diclofenaco de sódio 50mg, a cada oito horas de acordo com a dor.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Os pacientes selecionados foram alocados de forma aleatória através da lista de randomização gerada por computador, foram confeccionados envelopes lacrados e opacos utilizados para manter o segredo de alocação. Todos foram submetidos à avaliação inicial (T0), com 20 dias (T20) e com 45 dias (T45), por um avaliador cego.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy treatment technique (Experimental): Randomized clinical trial controlling and using at the time of allocation, toss with sealed envelopes, sealed and opaque. The study group will be dealt with "technical isostretching"
  Interventions: Other: Isostretching
- Patients remained on the waiting list (No Intervention): Randomized clinical trial controlling and using at the time of allocation, toss with sealed envelopes, sealed and opaque. The study group will be dealt with control group.

INTERVENTIONS:
Other: Isostretching — 12 interventions (two times per week) for 45 minutes
  Other Names: Strengthening and stretching exercise during expiration.
  Arms: Physiotherapy treatment technique

SUMMARY:
Isostretching is effective in treating chronic back pain to improve pain, quality of life and functional capacity.

DETAILED DESCRIPTION:
Objective: This study investigated the influence of isostretching on patients with chronic low back pain. Methods: It was a randomized, controlled trial with concealed allocation, intention-to-treat analysis, and blind assessment. Fifty-four patients with chronic low back pain were randomized to an experimental group and a control group. The experimental group performed isostretching twice a week for 45 days, while the control group remained on the waiting list for physical therapy. Patients were submitted to evaluations at baseline, after 20 and 45 days of treatment with regard to pain, quality of life, functional capacity, and satisfaction. Results: The experimental group exhibited statistically significant improvements in comparison to the control group with regard to pain (p = .003), functional capacity (p = .026), patient satisfaction (p < .001), and quality of life as determined by the functional capacity (p = .012), physical aspects (p = .011) and pain (p = .006) subscales of the SF-36. The experimental group used a significantly lesser amount of pain medication than the control group (p = .03). Conclusion: Isostretching was effective in reducing pain and in improving function, patient satisfaction and some aspects of quality of life in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic low back pain with pain located between the last rib and the gluteal fold over 12 weeks;
* Mechanical back pain that worsens with exertion and relieved by rest;
* Pain between 3 and 8 cm measured by analog pain scale.

Exclusion Criteria:

* Subjects who presented pain root
* Fibromyalgia
* Severe scoliosis with abnormal alignment of the spine (Cobb angle> 40); Tumors in the column; Infiltration in the lumbar spine in the last three months; Previous surgery of the spine (patients return to work or process expulsion)
* Have changed or initiated physical activity in the last three months
* Body mass index greater than 30 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of isostretching effects in patients with chronic low back pain | 1 month
  Reviewed by analog pain scale. (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Rosângela A Prado, Specialist, Principal Investigator — Universidade Estadual de Ciências da Saúde de Alagoas
Locations (1):
- Erika Rosangela Alves Prado, Maceió, Alagoas, Brazil